CLINICAL TRIAL: NCT02865863
Title: Safety and Efficacy Profile of the Eurycomalongifoliawaterextract (Physta®)+Multivitamin Study Product
Brief Title: A Study to Evaluate the Effect of a Study Product on Quality of Life and Mood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Biotropics Malaysia Berhad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BIOT2600
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Quality of Life; Mood
Keywords: Multivitamin; Eurycomalongifoliawater extract; Quality of Life; Mood
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Eurycomalongifoliawater extract (Physta®) +Multivitamin (Experimental)
  Interventions: Dietary Supplement: Eurycomalongifoliawater extract (Physta®); Dietary Supplement: Multivitamin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Eurycomalongifoliawater extract (Physta®)
  Arms: Eurycomalongifoliawater extract (Physta®) +Multivitamin
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Multivitamin
  Arms: Eurycomalongifoliawater extract (Physta®) +Multivitamin

SUMMARY:
A phase II randomized, placebo controlled study evaluating the efficacy of Eurycomalongifoliawater extract (Physta®)+Multivitamin on quality of life and mood on 86 healthy adults over a 24 week supplementation period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects ≥ 25 and ≤ 65 years of age.
* Body mass index (BMI) ≥ 18 and ≤30 kg/m2.
* Subjects must be employed in a job/position that has some degree of responsibility such that they experience a mid-level of stress at work.
* Subjects with a score of ≤ 18 in the Tension subscale and a score of ≤ 14 in the Fatigue subscale of the POMS Questionnaire.
* Judged by the Investigator to be in general good health on the basis of medical history.
* Females of child-bearing potential must agree to use appropriate birth control methods during the study.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator

Exclusion Criteria:

* Subjects with any history of immune system disorder or auto-immune disorder including but not limited to the following:

  *AIDS, HIV, Ankylosing Spondylitis, Chronic Fatigue Syndrome, CREST syndrome, Crohn's disease, Dermatomyositis, Fibromyalgia, Grave's disease, Hashimoto's Thyroiditis, Lupus, Multiple Sclerosis, Myasthenia Gravis, Pernicious Anemia, PolyarteritisNodosa, Primary Biliary Cirrhosis, Psoriasis, Reynaud's Syndrome, Rhematoid Arthritis, Sarcoidosis, Scleroderma, Sjogren's Syndrome, Temporal Arthritis, Ulcerative Colitis, and Vitiligo
* Use of any immunosuppressive drugs in the last 12 months (including steroids or biologics)
* Any significant GI condition that would severely interfere with the evaluation of the study product including but not limited to inflammatory bowel disease (Ulcerative Colitis or Chron's), history of frequent diarrhea, history of surgery for weight loss (including gastric bypass or lapband), history of perforation of the stomach or intestines, gastroparesis, clinically important lactose intolerance
* Any active infection, or infection in the last month requiring antibiotics, antiviral medication, or hospitalization History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Subjects with a history of seizure
* Recent history of (within 12 months) or strong potential for alcohol or substance abuse.
* Participation in a clinical study with exposure to any non-registered drug product within 30 days prior.
* Subject who are using herbal products containing androgenic/anxiolytic activity within 30 days (one month washout is allowed)
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk. Including subjects who are Bed or wheelchair-bound
* Untreated or unstable Hypothyroidism
* Subjects with active eating disorder including anorexia nervosa, bulimia, and/or obsessive compulsive eating disorders
* Central Neurological disorders including but not limited to Spinal cord injuries, multiple sclerosis, Parkinson's disease
* Pregnant, lactating, planning to become pregnant or unwilling to use adequate contraception during the duration of the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The change in quality of life after 24 weeks of supplementation with study product, measured using the SF-12 Quality of Life Questionnaire | 24 Week
The change in mood after 24 weeks of supplementation with study product, measured using the POMS Questionnaire | 24 week

SECONDARY OUTCOMES:
The change in stress after 24 weeks of supplementation with study product, measured using the Multi-Modal Stress Questionnaire | 24 weeks
The change in fasting AM Cortisol levels after 24 weeks of supplementation with study product. | 24 weeks

OTHER OUTCOMES:
The change in CBC levels after 24 weeks of supplementation with study product | 24 weeks
The change in CMP results after 24 weeks of supplementation with study product | 24 weeks
The change in urinalysis results after 24 weeks of supplementation with study product | 24 weeks
The number of adverse events reported after 24 weeks of supplementation with study product | 24 weeks
The change in lipid panel results after 24 weeks of supplementation with study product | 24 weeks
The change in total testosterone results after 24 weeks of supplementation with study product | 24 weeks
The change in free testosterone results after 24 weeks of supplementation with study product | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: TengkuShahrirTengku Adnan, Study Director — Biotropics Malaysia Berhad

REFERENCES:
- [Derived] George A, Udani J, Abidin NZ, Yusof A. Efficacy and safety of Eurycoma longifolia (Physta(R)) water extract plus multivitamins on quality of life, mood and stress: a randomized placebo-controlled and parallel study. Food Nutr Res. 2018 Oct 16;62. doi: 10.29219/fnr.v62.1374. eCollection 2018. PMID 30574050